CLINICAL TRIAL: NCT04074694
Title: Treatment of Juvenile Recurrent Parotitis: the Yield of Minimally Invasive Intervention, a Prospective Controlled Study
Brief Title: Treatment of Juvenile Recurrent Parotitis: the Yield of Minimally Invasive Intervention
Acronym: JRP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Carmel Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMC-18-0075-CTIL
Record Dates: First submitted 2019-08-29; First posted 2019-08-30 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Parotitis, Juvenile Recurrent
Keywords: Parotitis; Juvenile; Sialoendoscopy; Watchfull waiting
MeSH Terms: conditions — Parotitis, Juvenile Recurrent; Parotitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Watchfull waiting (No Intervention)
- Interventional (Active Comparator)
  Interventions: Procedure: Sialoendoscopy

INTERVENTIONS:
Procedure: Sialoendoscopy — Sialoendoscopy
  Arms: Interventional

SUMMARY:
Juvenile recurrent parotitis (JRP) is an inflammatory disease characterized by recurrent painful swelling of the Parotid gland in the pediatric age. A watchful waiting treatment strategy was acceptable for most children; however, recent studies claimed that a sialoendoscopic intervention may stop the recurrent flare-ups.

The Objective of our study:

To determine the effectiveness of sialoendoscopy vs. conservative therapy ('watch and wait') alone for Juvenile Recurrent Parotitis

Research Endpoints:

The study's endpoints will evaluate frequency and severity of flare-ups before and after treatment and Quality of Life parameters as evaluated according to life-quality questionnaires.

DETAILED DESCRIPTION:
Juvenile recurrent parotitis (JRP) is an inflammatory disease characterized by recurrent painful swelling of the Parotid gland in the pediatric age. A watchful waiting treatment strategy was acceptable for most children; however, recent studies claimed that a sialoendoscopic intervention may stop the recurrent flare-ups.

Moreover, the accessibility to this treatment modality and furthermore to the skillful operators are yet limited in many medical centers.

Juvenile Recurrent Parotitis is defined as a non-obstructive, non-suppurative inflammatory disease characterized by unilateral or bilateral parotid gland swelling recurring at least twice before puberty. It is the second most common salivary gland disease in children after mumps, in young children it is difficult to differentiate between the two. The clinical symptoms of JRP include intermittent and usually unilateral (might also be bilateral, usually with symptoms more prominent on one side) swelling of the parotid gland which occurs in quite a sudden pattern (over a course of houres or even minutes) and may persist for days or weeks, usually associated with local pain and erythema of the overlying skin, and systemic manifestation such as malaise and fever. The first episode typically occurs between ages 3-6, more often in males than females.

The etiology of JRP is still obscure, though a variety of causative factors have been proposed as contributing to JRP, such as dental congenital malformations, congenital duct malformation, genetic factors and immunological anomalies.

In addition to the conservative follow-up treatment modality, management with operative endoscopic treatment is another considerable option, that is now gaining stronger evidence of efficacy.

The procedure of sialoendoscopy has an increasing value of diagnosis and treatment of JRP, as it provides direct visualization of the ductal system and the abilty of treatment via lavage and irrigation of medical agents, such as steroids. There are a few reports indicating better outcomes (e.g. fewer exacerbations) using this modality

The Objective of our study:

To determine the effectiveness of sialoendoscopy vs. conservative therapy ('watch and wait') alone for Juvenile Recurrent Parotitis

Research Endpoints:

The study's endpoints will evaluate frequency and severity of flare-ups before and after treatment and Quality of Life parameters as evaluated according to life-quality questionnaires.

Inclusion criteria:

* age 3-18 y/o
* at least 2 documented incidents in at least 12 months period

Exclusion criteia:

* previous parotis interventions e.g. sialography/sialendoscopy/parotidectomy
* parotitis due to any other known cause (e.g. bacterial infection, autoimmune disease etc.)

ELIGIBILITY:
Inclusion Criteria:

age 3-18 y/o at least 2 documented incidents in at least 12 months period

Exclusion Criteria:

previous parotis interventions e.g. sialography/sialendoscopy/parotidectomy parotitis due to any other known cause (e.g. bacterial infection, autoimmune disease etc.)

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of flare-ups | 3 years
Quality of Life (QoL ) Questionnaire | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Otolaryngology, Carmel Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No